CLINICAL TRIAL: NCT05523505
Title: Bridging the Gap Between Brain Network Science and High-definition Non-invasive Brain Stimulation to Develop a Scalable Adult Literacy Intervention
Brief Title: Noninvasive Brain Stimulation to Enhance Reading Comprehension Ability in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Katherine Aboud, Research Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 220596; DP5OD031843 (NIH)
Record Dates: First submitted 2022-08-17; First posted 2022-08-31 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Reading Disability
Keywords: Neuroimaging; Adults; Non-invasive Brain Stimulation; Reading; Reading Comprehension
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Sham stimulation (Sham Comparator): Participants receiving sham stimulation.
  Interventions: Device: Sham intervention
- Reading and Language Network (RLN) (Experimental): Participants receiving real stimulation to the left angular gyrus.
  Interventions: Device: RLN real non-invasive brain stimulation intervention
- RLN and CCN (Experimental): Participants receiving real stimulation to the left dorsolateral prefrontal cortex and left angular gyrus.
  Interventions: Device: RLN and CCN real non-invasive brain stimulation intervention

INTERVENTIONS:
Device: Sham intervention — Use of the non-invasive brain stimulation device to simulate peripheral experience of stimulation without actually stimulating the brain.
  Arms: Sham stimulation
Device: RLN real non-invasive brain stimulation intervention — Real non-invasive brain stimulation to the left angular gyrus using transcranial alternating current stimulation (tACS).
  Arms: Reading and Language Network (RLN)
Device: RLN and CCN real non-invasive brain stimulation intervention — Real non-invasive brain stimulation to the left dorsolateral prefrontal cortex and left angular gyrus using transcranial alternating current stimulation (tACS).
  Arms: RLN and CCN

SUMMARY:
The goal of this project is to address the urgent need for effective, scalable adult literacy interventions by integrating breakthroughs in two separate fields: 1.) the brain network science of resilience to reading disorders and 2.) high-definition non-invasive brain network stimulation. This study will first establish the efficacy of a novel, noninvasive stimulation protocol on reading behavior and brain metrics; then will determine how stimulation-induced effects interact with baseline reading comprehension ability; and lastly, will identify whether stimulation-induced effects are more clinically-beneficial than canonical behavioral interventions. Results may change the foundation for how we treat low adult literacy, and have the potential for wider reaching impacts on non-invasive stimulation protocols for other clinical disorders.

DETAILED DESCRIPTION:
One in five adults in the US are unable to adequately comprehend a sentence. Low literacy is a major public health crisis, with no existing solution: findings from the Programme for the International Assessment of Adult Competencies (PIAAC) reveal that there have been no significant improvements to US national statistics on literacy in the past 30 years. Studies of the survey data reveal that adults with low literacy in the US have in-tact but slow word reading processes and vocabulary, and struggle to comprehend sentences and passages. Rates of poor reading comprehension (RC) ability are especially alarming given that RC ability is strongly predictive of educational outcomes, occupation and wage, health literacy/outcomes, and crime. Through these links, the World Literacy Foundation estimates that the literacy crisis accounts for 2% of the US's GDP annually. The current gold-standard interventions for RC ability are behavioral interventions that focus on cognitive skills found to support RC. However, meta-analyses across interventions show minimal raw gains. Brain research has allowed for the identification of "hidden" RC processes that are not captured by behavioral tests These studies have identified a consistent brain pathway that supports positive RC outcomes. This pathway is a compelling target for brain-based interventions. In particular, recent advances in noninvasive brain stimulation interventions provide a promising route for clinically-meaningful, brain-based treatments. However, brain research in RC has not been translated into an effective brain-based intervention. There is an urgent need for a cutting-edge, non-invasive brain stimulation intervention that will transform the way we approach the clinical treatment of poor RC. The current project will integrate our work in the brain network science of RC and breakthroughs in non-invasive stimulation to address these challenges and develop a brain-based RC intervention.

To accomplish this, the proposed study will invite typical adults with a range of RC ability (good and poor) to participate in three visits to the lab. The rationale for examining adults is to that the current study aims to develop a brain-based intervention (i.e. non-invasive brain stimulation) to treat low literacy in adults, as current behavioral interventions in adults are largely unsuccessful. N=100 participants will come in for three visits; for each visit adults will complete behavioral testing, magnet resonance imaging (MRI), and electroencephalography (EEG). Visit 1 will establish baseline behavior and brain measures of the individual (total visit time of 3.5 hours). Visit 2 will include a behavioral and safe, non-invasive stimulation intervention for the individual (total visit of 3 hours). Stimulation will involve two sessions, one while subjects are in the MRI, and one while subjects are having EEG. Visit 2 will also involve behavioral testing to determine intervention effects. Visit 3 will establish prolonged intervention effects using behavior and brain measures of the individual (total visit of 2.5 hours). Participants will be recruited and randomly assigned to receive one of three non-invasive stimulation interventions, and all will receive a canonical behavioral intervention, so that the smallest subgroup in the study will be N=30, which provides sufficient statistical power (see Statistical Design and Power). All subjects will have typical word reading ability (greater than or equal to 15th percentile), and either good (greater than 25th percentile) or poor (less than or equal to 25th percentile) reading comprehension ability. Non-invasive stimulation subgroups include two stimulation groups distinguished only by electrode placement, and one sham control group. Behavioral intervention involves a short paper/pencil reading comprehension intervention. Each intervention subgroup will be randomly assigned, but with the restriction that the distribution of reading comprehension ability is even across subgroups. This will be accomplished while maintaining double-blind procedures. Collection will begin in Summer 2022 and continue through Fall 2026. Adults will be recruited from the Nashville community. Behavioral testing and MRI (with and without stimulation) will occur at the Vanderbilt Institute for Imaging Science (VUIIS). EEG (with and without stimulation) will occur at the Vanderbilt Kennedy Center.

ELIGIBILITY:
Inclusion Criteria:

This study will be open to all right-handed, native English monolingual speakers, who meet eligibility criteria regardless of race, gender, minority or socioeconomic status. Due to age-related differences in the language and learning processes, the age range of subjects will be a minimum of 18 years and a maximum of 40 years.

Exclusion Criteria:

We will exclude individuals with a personal medical history of stroke or seizures or those taking medications specifically prescribed for the treatment of stroke or seizures. However, participants who are on medications that carry an associated risk of stroke or seizures but are not prescribed for these conditions (e.g., anticonvulsants prescribed for pain or behavioral reasons) will remain eligible. Exclusion criteria will be determined by follow-up telephone screenings conducted by lab KSP and is as follows:

1. previous diagnosis of Intellectual Disability;
2. known uncorrectable visual impairment;
3. documented hearing impairment greater than or equal to a 25 dB loss;
4. medical contraindication to MRI procedures (e.g., metal devices);
5. known IQ below 70;
6. a pervasive developmental disorder;
7. any known neurologic pathology, including epilepsy, spina bifida, cerebral palsy, traumatic brain injury, and brain tumors;
8. recent medical diagnosis of migraines;
9. pregnancy;
10. history of syncope;
11. severe fatigue,
12. bilingualism or low English proficiency;
13. poor reading ability that will prevent completion of the tasks; and
14. comorbid severe psychiatric disorders will be excluded;
15. a personal medical history of stroke or seizures;
16. hair styles that do not allow for proper EEG net fitting, or that pose potential risks for damage to EEG net

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in reading comprehension ability on standardized test measure | Baseline to 12 months
  Stimulation induced change in reading comprehension ability measured by Gates MacGinitie Reading Test:
  * Reading Comprehension Subtest (Adult Reader; AR): Participants have 35 minutes to read passages and answer 48 comprehension questions about what they read.
  * Percentile Ranks based on the scores of entering community college students
  * Primary outcome measure is the change in percentile ranks
Performance in reading comprehension ability on test measure during stimulation session | Baseline to 12 months
  Stimulation induced performance in reading comprehension ability measured by free recall of information learned while reading during stimulation session.
  * Subject asks to recall content from 100 total sentences
  * Primary outcome measure is the number correct out of total (# recalled / total) compared across groups (real stimulation subgroups and sham).

SECONDARY OUTCOMES:
Change in brain activations during reading | Baseline to 12 month
  Stimulation induced change in brain activations during reading as measured by a joint analysis of functional magnetic resonance imaging and electroencephalography.
  * Measures of co-activation in brain areas are obtained for certain timepoints during sentence reading.
  * Typical brain patterns over time are obtained from readers without reading difficulties.
  * The primary outcome measure is a weighting value that reflects how strongly a subject's brain signals align with expected brain signals for typical reading processes.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine S. Aboud, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
All research resources and other information developed in this project will be made readily available to the scientific community to support replication of the study's research findings as well as big-data initiatives. Anonymized raw neuroimaging data, demographic data (including age, sex, ethnicity, handedness, and socioeconomic status), and neuroimaging collection parameters will be deposited in the open source data base, NITRC (NeuroImaging Tools and Resources Collaboratory). This will be made publicly available within six months of the initial publication of the data, which we anticipate will occur in year 5 of the proposed research. Other mechanisms for the transfer of information, including research findings and relevant code, will take the form of peer-reviewed publications with links to open source code, posters at scientific conferences and research presentations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available no more than 6 months after initial publication.
Access Criteria: Publicly available.

DOCUMENTS (1):
  • Informed Consent Form (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT05523505/ICF_000.pdf